CLINICAL TRIAL: NCT05380089
Title: Effects of Hydration Changes on Neuromuscular Function of Athletes With Low Water Intake
Brief Title: Effects of Hydration Changes on Neuromuscular Function of Athletes
Acronym: H2OAthletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H2O Athletes
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Dehydration; Hyperhydration
Keywords: Electromyography; hydration status; neuromuscular activation; muscle strength; muscle power; hydration assessment; dehydration; body composition
MeSH Terms: conditions — Dehydration; Water Intoxication

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial (RCT)
Masking Description: Given the nature of the study, it is not possible to blind neither participants nor research team members regarding the allocated groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Over a 4-day period, participants randomly assigned to the experimental group will be instructed to maintain normal solid food choices, but to increase water intake to achieve a total water intake of ≥45ml/kg/day. Prepared bottles of water with the required amount will be given to each participant every morning and collected empty the following day. Instructions to drink small amounts of water every hour be transmitted.
  Adherence to instructions regarding water intake will be determined by the return of drinking bottles, analysis of daily food records, assessment of water flux (i.e., collecting urines after subjects being dosed with deuterium), and daily screening questions. These samples will be delivered on a subsequent morning during a daily laboratory visit to collect urine and saliva samples, as well as BI assessment. On the 4th day, participants will perform a neuromuscular function assessment.
  Interventions: Other: Increasing water intake
- Control group (No Intervention): Participants randomly assigned to the control group will be instructed to maintain normal solid food choices and water intake based on their average intake reported on the food records. Adherence to instructions regarding water intake will be determined and assessments performed will occur as mentioned previously for the experimental group.

INTERVENTIONS:
Other: Increasing water intake — Participants randomly assigned to the experimental group will be instructed to maintain habitual solid food choices and to increase water intake to achieve a total water intake of ≥45ml/kg/day.
  Arms: Experimental group

SUMMARY:
Greater muscular strength and power are relevant qualities for athletic success and decreased injury rate. It is known that dehydration impairs muscular strength and power, although the explanation for this association is not entirely clear. Besides morphological factors, strength production also depends on neural factors which in turn can be affected by dehydration. Some studies tested the effects of dehydration on neuromuscular function using electromyography (EMG) analysis. However, there is no consensus among those studies.

Additionally, exercise may disturb water balance. This can further lead to dehydration if the athlete does not properly rehydrate. In this sense, the scientific evidence has identified people who are considered low drinkers that may be more susceptible to cellular shrinkage, potentially impairing health and performance. Thus, it would be expected that athletes regularly exposed to lower amounts of water intake would have beneficial effects in both performance and health if higher water ingestion was promoted, namely an improved neuromuscular function via enhanced cellular hydration. However, any potential benefit of increasing water intake on neuromuscular function is still to be determined using well-designed experimental studies and state-of-the-art methods.

Lastly, there is no consensus regarding the diagnosis of dehydration in athletes. The identification of simple indices to measure dehydration in athletes is crucial as many may be inaccurately diagnosed.

DETAILED DESCRIPTION:
Athletes are dependent on muscular strength as it is associated with a higher rate of force development and muscular power, general and specific sports skills performance, and decreased injury rates. There is scientific evidence showing that a hypohydrated state [i.e., 2 to 3% of body mass loss (BML) attributed to water loss] impairs muscular strength and power. However, how this reduction affects athletic performance remains in question.

We know that muscular strength development is derived from a combination of morphological (muscle cross-sectional area, muscle architecture, and musculotendinous stiffness) and neural factors (motor unit recruitment, synchronization, and firing frequency). Thus, neural factors may be one possible explanation for the effects of dehydration. In fact, there is biological plausibility for this relation as dehydration may affect the electrolyte's concentration (particularly potassium and sodium) within intra- and extracellular spaces, leading to an alteration of the membrane electrochemical potential.

Although some studies have tested the effects of hydration changes on neuromuscular function using electromyography (EMG) analysis, there is still no consensus among them. Some authors showed effects of dehydration on muscle endurance and EMG signal, including reduction in EMG mean power frequency (MPF) and an accelerated rate of root-mean square (RMS), possibly meaning reduced membrane excitability and an accelerated central mediated regulation of motor unit activity. While others did not find any effect of dehydration on EMG values. Thus, experimental studies using well-designed trials and state-of-the-art technology are required to better understand the effects of acute dehydration on neuromuscular function, specifically in athletes.

Maintenance of a euhydrated state is crucial for the proper physiological functioning of the body, being achieved by physiological and behavioral factors. However, exercise can disturb water balance, particularly when performed in hot environments, increasing water loss. This can further lead to dehydration if the athlete does not properly rehydrate. In this sense, the scientific evidence has identified people who are considered low drinkers (i.e., people who are exposed to a low regular water intake) and high drinkers (i.e., people who are exposed to a high regular water intake). These differences in water intake lead to different physiological responses such as serum arginine vasopressin (AVP) levels and also in mood states. Although no specific total water intake guidelines have been established for athletes, when compared to the European Food Safety Authority guidelines for water intake in healthy adults, they do not meet the guidelines, specifically when higher hydration needs are considered. As mentioned before, AVP has been used to distinguish low drinkers from high drinkers, namely elevated plasma AVP in low drinkers suggesting intracellular dehydration.

In fact, changes in total body water (TBW) and its compartments [i.e., intracellular water (ICW) and the extracellular water (ECW)] have been studied regarding their impact on sports performance. Silva and colleagues observed that judo athletes who decrease TBW, namely by decreasing ICW, were those that decreased upper-body power, regardless of changes in weight and arms' lean-soft tissue. Also, ICW was the only body water compartment whose reductions explained the higher probability of losing >2% of forearm maximal strength, independently of changes in weight and arms' lean-soft tissue. Finally, ICW was also considered the main predictor of strength and jumping height over the season in national-level athletes. Thus, ICW and cellular hydration appear to play a relevant role in athletic power and strength, although further research is needed to link these structural fluid compartments with changes in the hydration status and its connection with neuromuscular function.

Lastly, hydration testing has been considered a controversial topic and despite existing a substantial body of research, there is no clear protocol regarding the best practice for assessing hydration status in athletes. Moreover, new methods that provide hydration status safely, accurately, reliably, and feasibly are also needed. Bioelectrical Impedance Analysis (BI) is an alternative technique for this specific context. The BI method utilizes the components of impedance: resistance (R) and reactance (Xc). Phase angle (PhA) is also provided, representing a relevant indicator of cellular health and muscle functionality, but research is lacking on the usefulness of this marker for tracking strength/power in athletes exposed to short-term changes in hydration status.

To summarize, there is a lack of evidence-based protocols with the state-of-the-art methodology to test the effects of modifying water intake on neuromuscular function using EMG analysis in the athletic population. Moreover, the currently available experimental designs present methodological limitations in assessing hydration status and body water compartments. Hence, to overcome the shortcomings, innovative research with cutting-edge technology is required. Thus, our primary aim is to determine the effects of hydration changes (i.e., a 4-day intervention targeting raises in water intake and acute dehydration) on the strength and power (with EMG analysis for the neuromuscular response) of athletes. Secondary aims include: i) to compare the effects of acute dehydration on neuromuscular function before and after the intervention; ii) to analyze the effects of the intervention on TBW, ECW, ICW, and fat-free mass (FFM) hydration; iii) to analyze the effects of hydration changes (I.e., a 4-day intervention targeting raises in water intake and acute dehydration) on several hydration indexes (serum, saliva, and urine osmolality) and biochemical markers (AVP and sodium concentration); iv) to test the usefulness of segmental and whole-body raw BI parameters in detecting acute dehydration using serum osmolality as the reference technique; v) to explore if PhA can be used as a marker of neuromuscular function;

ELIGIBILITY:
Inclusion Criteria:

* Highly trained athletes (i.e., participating in national and international championships and/or ≥6 h of training per week)
* Athletes considered low drinkers (i.e., total water intake ≤ 35ml/kg/)
* Aged between 18 and 35 years
* Living in Lisbon and/or its surroundings
* All women should have a (self-reported) normal menstrual cycle (i.e., cycles at median intervals of less than 35 days)
* Completion of the sport's medical examination

Exclusion Criteria:

* Total water intake above 35ml/kg/day.
* Clinical history compatible with exertional heat illness (i.e., heat stroke, heat exhaustion, hyperthermia, among other events that suggest poor response to thermically challenging environments)
* Taking medication known to alter the normal fluid-electrolyte balance, plasma osmolality, urinary osmolality, or the chronotropic response to exercise (e.g., diuretics, antidiuretics, laxatives, oral contraceptives, drugs to control blood pressure (39)
* Exhibiting self-reported metabolic disorders or malfunction of salivary glands
* Active smoking status
* Unwilling to abstain from alcohol during this study
* Respiratory disorders, including asthma
* Injuries that would limit exercise performance
* Mechanical prostheses
* Pregnancy /planning to get pregnant within the next 8 months
* Having been pregnant within the past 6 months or breastfeeding
* Failure to complete the dietary intake and physical activity recording
* Unable to communicate with local study staff
* Needle phobia
* Inability to complete the study within the designated time frame because of plans to move out of the study area or occurrence of competition periods during the study timeframe
* Inability to attend the visits/appointments and evaluation measurements

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum voluntary isometric contraction - Knee extension | 3 weeks
  For the lower body strength, participants will be assessed on a Biodex System 3 Pro isokinetic dynamometer (Biodex Medical Systems, Shirley, NY). The participants will remain seated with the belts positioned on the thorax, abdomen, thigh, and above the knee on the side that is being evaluated to limit the knee movement.
  Each testing session will begin with a dynamic warm-up, consisting of 5min of submaximal cycle-ergometry set at 25 W followed by a 5 min of resting before starting the testing protocol. First, a MVIC 5-s voluntary knee extension (knee at 70o for the extension). Verbal encouragement and audible feedback from the dynamometer software will be provided to each participant.
Maximum voluntary isometric contraction - Knee flexion | 3 weeks
  After the maximum voluntary isometric contraction for knee extension, participants will be asked to perform a MVIC 5-s voluntary knee flexion (30o for the flexion). This test will be performed with 3min of pause after the MVIC of knee extension.
Rate of torque development (RTD) for knee extension and flexion | 3 weeks
  In both MVIC for knee extension and flexion, the participants will be instructed to avoid any countermovement prior to test and will be asked to exert their maximum force as fast and hard as possible, to obtain both maximal torque and rate of torque development (RTD). Verbal encouragement and audible feedback from the dynamometer software will be provided to each participant.
5 submaximal isometric repetitions of knee extension | 3 weeks
  5 submaximal isometric repetitions will me measuredfrom MVIC of baseline and MVIC of that day: 1) 30s at 20% of MVIC; 2) 30s at 40% of MVIC; 3) 10s at 60% of MVIC; 4) 10s at 80% of MVIC; 5) 10s at 100% of MVIC. Between repetitions a pause of 1 min will be performed between repetitions while a pause of 3 min will be performed between sets.
Fatigue task | 3 weeks
  Last, and after a pause of 5 min, participants will perform an isometric contraction at 40% of MVIC (measured on the day) until to exhaustion. Exhaustion will be considered if a decrease of more than 10% of MVIC for more than 10s is observed.
EMG signals - Root mean square | 3 weeks
  During the legs' strength assessment, EMG signals will be recorded (EMG Delsys Trigno Avanti, Delsys Incorporated, USA) from the vastus lateralis (VL), rectus femoris (RF), vastus medialis (VM), and biceps femoris (BF) muscles in accordance with the guidelines of the Surface EMG for the Non-invasive Assessment of Muscles (SENIAM). The electrodes will be placed before the 5 min of resting after the dynamic warm-up. EMG signals from each muscle will be pre-amplified (gain 1000), band-pass filtered (20-450 Hz), and A/D converted at 1kHz (MP100, BIOPAC Systems Inc., Goleta, CA). AcqKnowledge 4.3.1 software will be used for data collection and processing (BIOPAC Systems Inc., Goleta, CA).
EMG signals - Mean power frequency | 3 weeks
  During the legs' strength assessment, EMG signals will be recorded (EMG Delsys Trigno Avanti, Delsys Incorporated, USA) from the vastus lateralis (VL), rectus femoris (RF), vastus medialis (VM), and biceps femoris (BF) muscles in accordance with the guidelines of the Surface EMG for the Non-invasive Assessment of Muscles (SENIAM). The electrodes will be placed before the 5 min of resting after the dynamic warm-up. EMG signals from each muscle will be pre-amplified (gain 1000), band-pass filtered (20-450 Hz), and A/D converted at 1kHz (MP100, BIOPAC Systems Inc., Goleta, CA). AcqKnowledge 4.3.1 software will be used for data collection and processing (BIOPAC Systems Inc., Goleta, CA).
Handgrip strength | 3 weeks
  The handgrip strength test measures maximum voluntary isometric contraction (MVIC) of the hand and forearm muscles. Handgrip will be performed using a portable hand dynamometer (TSD121C; Biopac Systems, Goleta, CA, USA). Participants will be assessed on both hands alternately, in a standing position. Prior to the test, the grip dynamometer will be adjusted to the size of the hand of each subject. Handgrip strength assessment will be conducted with the subject standing up with the arms in a neutral position (halfway between supine and pronation position). Each participant will be assessed on both hands alternately until reaching 3 attempts for each hand. In each attempt, the subject will exert the maximal grip strength on the handgrip dynamometer with the assessed hand for 5s. After each attempt, there will be a resting period of 60s that will be used both for recovery and for changing the handgrip dynamometer to the opposite hand.

SECONDARY OUTCOMES:
Food records | 3 weeks
  A trained dietitian will calculate the athlete's habitual total water intake (i.e., the sum of the water present in beverages and the water in foods) based on a 3 non-consecutive days food record. Before filling the food records, a registered dietitian will provide written instructions using specific guidelines, pictures of portion sizes, and examples of common errors in recording dietary intake. The Portuguese Food guide will be used for the estimation of ingested portions. For the conversion of the contribution of water from food, the software package Food Processor Plus® (ESHA Research, USA) will be used by a registered dietitian.
Cardiorespiratory Fitness Test | 3 weeks
  A trained exercise physiologist will perform a maximal cardiorespiratory fitness test using an incremental test on variable speed and incline treadmill (Pulsar 3p, HP Cosmos, Nussdorf-Traunstein, Germany).The participants will perform the incremental test until exhaustion to determine their VO2max and the VT. The test will start with a 5-min seated period followed by a 1-min warm-up at 8kmh-1 with consecutive increases of 1kmh-1 per minute until exhaustion. Recovery consisted of a 3 min walk at 2.4kmh-1 speed and a grade of 2.5%.
  Expired gas measurements will be taken using a breath-by-breath metabolic cart (QUARK RMR, version 9.1, Cosmed, Rome, Italy). The VO2 and heart rate data, obtained throughout the graded exercise test, will be displayed in 20-s averages. The highest VO2 attained at the end of the test will be accepted as VO2max if a plateau in VO2 with an increase in treadmill speed was observed.
Plasma osmolality | 3 weeks
  Plasma osmolality (mOsm/kg) will be assessed by using the osmometer (Mod OSMO1, Advanced Instruments, Canada). Blood samples will be drawn from an antecubital vein via single venepuncture and will be collected in serum and plasma EDTA tubes. All blood samples will be centrifuged at 5000 rpm for 15 min at -4°C. Serum osmolality will be measured immediately following centrifugation.
Urine osmolality | 3 weeks
  Urine osmolality (mOsm/kg) will be assessed by using the osmometer (Mod OSMO1, Advanced Instruments, Canada). Urine osmolality (Uosm) is a measure of the number of dissolved particles per unit of water in urine. The osmolality of the urine sample reflects the self-regulating activity of renal concentration or dilution mechanisms during a 24-h period. Participants will receive a container for collecting and storing their urine.
  Blood samples will be drawn from an antecubital vein via single venepuncture and will be collected in serum and plasma EDTA tubes. All blood samples will be centrifuged at 5000 rpm for 15 min at -4°C. Serum osmolality will be measured immediately following centrifugation.
Saliva osmolality | 3 weeks
  Saliva (mOsm/kg) will be assessed by using the osmometer (Mod OSMO1, Advanced Instruments, Canada). For saliva sample collection, subjects then will provide unstimulated saliva by sitting quietly for 2min, allowing saliva to passively accumulate in the mouth. Then, participants will hold a salivette and remove its stopper. They will remove the swab from sallivete by tipping the container, so the swab falls directly into the mouth. To collect saliva, they will roll the swab in their mouth until they feel that they can no longer prevent their selves from swallowing the saliva produced. They will be instructed to not touch the swab with fingers during this process.
Thirst and mouth dryness | 3 weeks
  visual analogue rating scales of thirst and mouth dryness will be obtained. Participants will answer two questions by placing a mark on a 10 cm line according to their subjective analyses. The ends of the thirst line represent "Not at all thirsty" and "I'm very thirsty" and the question is "How thirsty do you feel now?". For mouth dryness the question is "How dry does your mouth feel now?" and the participants will mark the line between these ends representing "Not at all dry" and "Very dry".
Serum arginine vasopressin | 3 weeks
  Blood samples will be collected to assess serum AVP through ELISA.
Serum sodium concentration | 3 weeks
  Blood samples will be collected to assess serum sodium concentration by flame spectrometry
Total body water | 3 weeks
  Total body water (TBW) will be measured by deuterium dilution using a Hydra stable isotope ratio mass spectrometer (PDZ, Europa Scientific, UK). After a 12h fast, the first urine sample will be collected. Each participant will take an oral dose of 0.1g of 99.9% 2H2O per kg of body weight (Sigma-Aldrich;St. Louis, MO). After a 4h equilibration period, during which no food or beverage will be consumed, a urine sample will be collected as well as a urine sample at 5h. Urine and diluted dose samples will be prepared for 1H/2H analysis.
Extracellular water | 3 weeks
  Through the dilution of sodium bromide (NaBr), it will be possible the determination of ECW. After collection of a saliva sample, each participant will be asked to drink 0.030g of 99.0% NaBr (Sigma-Aldrich; St. Louis, MO) per kg of body weight, diluted in 50 mL of distilled deionized water. After a 3h equilibration period, during which no food or beverage will be consumed, a saliva sample will be collected. Saliva samples will be collected into salivettes. Then, the samples will be centrifuged and frozen for posterior analyses.
Intracellular water | 3 weeks
  Intracellular water (ICW) will be determined as the difference between TBW and ECW using the dilution techniques (ICW=TBW-ECW).
Phase angle | 3 weeks
  Whole body and segmental BI will be applied using the AKERN BIA 101/BIVA PRO, a phase-sensitive a single frequency bioelectrical impedance analysis (BIA) device that measures PhA.
Impedance | 3 weeks
  Whole body and segmental BI will be applied using the AKERN BIA 101/BIVA PRO, a phase-sensitive a single frequency bioelectrical impedance analysis (BIA) device that measures impedance (Z)
Resistance | 3 weeks
  Whole body and segmental BI will be applied using the AKERN BIA 101/BIVA PRO, a phase-sensitive a single frequency bioelectrical impedance analysis (BIA) device that measures PhA and impedance (Z), and then calculates resistance.
Reactance | 3 weeks
  Whole body and segmental BI will be applied using the AKERN BIA 101/BIVA PRO, a phase-sensitive a single frequency bioelectrical impedance analysis (BIA) device that measures PhA and impedance (Z), and then calculates reactance.
Classic Bioimpedance Vector Analysis (BIVA) | 3 weeks
  Classic BIVA will be performed, i.e., normalizing R and Xc parameters for stature (H) in meters. The length of the vector will be calculated as the hypotenuses of individual impedance values. The PhA will be calculated as the arc-tangent of Xc/R × 180°/π. Prior to each test, the analyser will be checked for calibration.
Fat mass | 3 weeks
  Fat mass (FM), a molecular component, is calculated from mathematical models, a reference 4-compartment model, as described below:
  FM (kg) = 2.748×BV - 0.699×TBW + 1.129×Mo - 2.051×BW, where BV is body volume (L) obtained by air displacement plethysmography (ADP, described below), TBW (kg) through dilution techniques (as described before), Mo is bone mineral (kg) obtained by dual-energy X-ray absorptiometry (DXA, described below), and BW is body weight (kg). Accordingly, FFM is calculated as FM minus BW. In this model soft minerals (Ms), a small molecular component, are calculated as 0.00129*TBW.
Body volume | 3 weeks
  Body volume will be assessed by ADP (BOD PODs, Life Measurement Inc., Concord, CA, USA). Each subject will wear a swimsuit and their body mass will be measured to the nearest 100g by an electronic scale connected to the plethysmograph computer. Body volume will be computed based on the initial BV corrected for thoracic gas volume and a surface area artifact computed automatically. The measured thoracic gas volume will be obtained in all subjects.
Bone mineral content | 3 weeks
  Bone mineral content will be estimated using DXA (Hologic Explorer-W, MA, USA). The attenuation of X-rays pulse between 70 and 140kV synchronously with the line frequency for each pixel of the scanned image. The lab technician will execute the analyses according to the operator's manual using the standard analysis protocol and considering the recommendations present in the literature. Considering that bone mineral content (BMC) represents ashed bone, BMC will be converted to total-body Mo by multiplying it by 1.0436.
Fat free mass | 3 weeks
  After the determination of FM, FFM is obtained by subtracting FM from body mass. As the main molecular components are determined, protein is also subtracted from FFM (Protein= FFM-TBW-Mo-Ms). The density of the FFM (FFMd) is also calculated as:
  FFMd = 1/((TBW/0.9937)+(Mo/2.982)+(Ms/3.317)+(Protein/1.34)) Thus, hydration of the FFM can be calculated as TBW/FFM. This value will be used as a reference to test the validity of the algorithm proposed in the AKERN BIA device.
Profile state of mood | 3 weeks
  The profile of mood states (POMS) questionnaire will be applied to assess distinct mood states. This questionnaire will be applied at baseline, before and after the dehydration protocols and after the 4-day intervention. The POMS is a 5-point self-administered scale that assesses various mood states.

CONTACTS AND LOCATIONS:
Overall Officials: Analiza Silva, PhD, Principal Investigator — Faculdade Motricidade Humana
Locations (1):
- Faculdade Motricidade Humana, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suchomel TJ, Nimphius S, Stone MH. The Importance of Muscular Strength in Athletic Performance. Sports Med. 2016 Oct;46(10):1419-49. doi: 10.1007/s40279-016-0486-0. PMID 26838985
- [Background] Judelson DA, Maresh CM, Anderson JM, Armstrong LE, Casa DJ, Kraemer WJ, Volek JS. Hydration and muscular performance: does fluid balance affect strength, power and high-intensity endurance? Sports Med. 2007;37(10):907-21. doi: 10.2165/00007256-200737100-00006. PMID 17887814
- [Background] Suchomel TJ, Nimphius S, Bellon CR, Stone MH. The Importance of Muscular Strength: Training Considerations. Sports Med. 2018 Apr;48(4):765-785. doi: 10.1007/s40279-018-0862-z. PMID 29372481
- [Background] Folland JP, Williams AG. The adaptations to strength training : morphological and neurological contributions to increased strength. Sports Med. 2007;37(2):145-68. doi: 10.2165/00007256-200737020-00004. PMID 17241104
- [Background] Casa DJ. Exercise in the heat. I. Fundamentals of thermal physiology, performance implications, and dehydration. J Athl Train. 1999 Jul;34(3):246-52. PMID 16558572
- [Background] Sjogaard G. Water and electrolyte fluxes during exercise and their relation to muscle fatigue. Acta Physiol Scand Suppl. 1986;556:129-36. PMID 3471050
- [Background] Barley OR, Chapman DW, Blazevich AJ, Abbiss CR. Acute Dehydration Impairs Endurance Without Modulating Neuromuscular Function. Front Physiol. 2018 Nov 2;9:1562. doi: 10.3389/fphys.2018.01562. eCollection 2018. PMID 30450056
- [Background] Ftaiti F, Grelot L, Coudreuse JM, Nicol C. Combined effect of heat stress, dehydration and exercise on neuromuscular function in humans. Eur J Appl Physiol. 2001 Jan-Feb;84(1-2):87-94. doi: 10.1007/s004210000339. PMID 11394259
- [Background] Evetovich TK, Boyd JC, Drake SM, Eschbach LC, Magal M, Soukup JT, Webster MJ, Whitehead MT, Weir JP. Effect of moderate dehydration on torque, electromyography, and mechanomyography. Muscle Nerve. 2002 Aug;26(2):225-31. doi: 10.1002/mus.10203. PMID 12210387
- [Background] Bigard AX, Sanchez H, Claveyrolas G, Martin S, Thimonier B, Arnaud MJ. Effects of dehydration and rehydration on EMG changes during fatiguing contractions. Med Sci Sports Exerc. 2001 Oct;33(10):1694-700. doi: 10.1097/00005768-200110000-00013. PMID 11581554
- [Background] Rodger A, Papies EK. "I don't just drink water for the sake of it": Understanding the influence of value, reward, self-identity and early life on water drinking behaviour. Food Quality and Preference. 2022;99:104576.
- [Background] Cheuvront SN, Kenefick RW. Dehydration: physiology, assessment, and performance effects. Compr Physiol. 2014 Jan;4(1):257-85. doi: 10.1002/cphy.c130017. PMID 24692140
- [Background] Belval LN, Hosokawa Y, Casa DJ, Adams WM, Armstrong LE, Baker LB, Burke L, Cheuvront S, Chiampas G, Gonzalez-Alonso J, Huggins RA, Kavouras SA, Lee EC, McDermott BP, Miller K, Schlader Z, Sims S, Stearns RL, Troyanos C, Wingo J. Practical Hydration Solutions for Sports. Nutrients. 2019 Jul 9;11(7):1550. doi: 10.3390/nu11071550. PMID 31324008
- [Background] Periard JD, Racinais S, Sawka MN. Adaptations and mechanisms of human heat acclimation: Applications for competitive athletes and sports. Scand J Med Sci Sports. 2015 Jun;25 Suppl 1:20-38. doi: 10.1111/sms.12408. PMID 25943654
- [Background] Perrier E, Vergne S, Klein A, Poupin M, Rondeau P, Le Bellego L, Armstrong LE, Lang F, Stookey J, Tack I. Hydration biomarkers in free-living adults with different levels of habitual fluid consumption. Br J Nutr. 2013 May;109(9):1678-87. doi: 10.1017/S0007114512003601. Epub 2012 Aug 31. PMID 22935250
- [Background] Armstrong LE, Munoz CX, Armstrong EM. Distinguishing Low and High Water Consumers-A Paradigm of Disease Risk. Nutrients. 2020 Mar 23;12(3):858. doi: 10.3390/nu12030858. PMID 32210168
- [Background] Johnson EC, Munoz CX, Le Bellego L, Klein A, Casa DJ, Maresh CM, Armstrong LE. Markers of the hydration process during fluid volume modification in women with habitual high or low daily fluid intakes. Eur J Appl Physiol. 2015 May;115(5):1067-74. doi: 10.1007/s00421-014-3088-2. Epub 2015 Jan 7. PMID 25564016
- [Background] Johnson EC, Munoz CX, Jimenez L, Le Bellego L, Kupchak BR, Kraemer WJ, Casa DJ, Maresh CM, Armstrong LE. Hormonal and Thirst Modulated Maintenance of Fluid Balance in Young Women with Different Levels of Habitual Fluid Consumption. Nutrients. 2016 May 18;8(5):302. doi: 10.3390/nu8050302. PMID 27213436
- [Background] Leiper JB, Pitsiladis Y, Maughan RJ. Comparison of water turnover rates in men undertaking prolonged cycling exercise and sedentary men. Int J Sports Med. 2001 Apr;22(3):181-5. doi: 10.1055/s-2001-15912. PMID 11354520
- [Background] Pross N, Demazieres A, Girard N, Barnouin R, Metzger D, Klein A, Perrier E, Guelinckx I. Effects of changes in water intake on mood of high and low drinkers. PLoS One. 2014 Apr 11;9(4):e94754. doi: 10.1371/journal.pone.0094754. eCollection 2014. PMID 24728141
- [Background] American College of Sports Medicine; Sawka MN, Burke LM, Eichner ER, Maughan RJ, Montain SJ, Stachenfeld NS. American College of Sports Medicine position stand. Exercise and fluid replacement. Med Sci Sports Exerc. 2007 Feb;39(2):377-90. doi: 10.1249/mss.0b013e31802ca597. PMID 17277604
- [Background] EFSA Panel on Dietetic Products N, Allergies. Scientific Opinion on Dietary Reference Values for water. EFSA Journal. 2010;8(3):1459.
- [Background] Nunes CL, Matias CN, Santos DA, Morgado JP, Monteiro CP, Sousa M, Minderico CS, Rocha PM, St-Onge MP, Sardinha LB, Silva AM. Characterization and Comparison of Nutritional Intake between Preparatory and Competitive Phase of Highly Trained Athletes. Medicina (Kaunas). 2018 May 30;54(3):41. doi: 10.3390/medicina54030041. PMID 30344272
- [Background] Pilis K, Stec K, Pilis A, Mroczek A, Michalski C, Pilis W. Body composition and nutrition of female athletes. Rocz Panstw Zakl Hig. 2019;70(3):243-251. doi: 10.32394/rpzh.2019.0074. PMID 31515983
- [Background] Nuccio RP, Barnes KA, Carter JM, Baker LB. Fluid Balance in Team Sport Athletes and the Effect of Hypohydration on Cognitive, Technical, and Physical Performance. Sports Med. 2017 Oct;47(10):1951-1982. doi: 10.1007/s40279-017-0738-7. PMID 28508338
- [Background] Arnaoutis G, Kavouras SA, Angelopoulou A, Skoulariki C, Bismpikou S, Mourtakos S, Sidossis LS. Fluid Balance During Training in Elite Young Athletes of Different Sports. J Strength Cond Res. 2015 Dec;29(12):3447-52. doi: 10.1519/JSC.0000000000000400. PMID 24513625
- [Background] Hall JE. Guyton and Hall textbook of medical physiology e-Book: Elsevier Health Sciences; 2015.
- [Background] Silva AM, Fields DA, Heymsfield SB, Sardinha LB. Body composition and power changes in elite judo athletes. Int J Sports Med. 2010 Oct;31(10):737-41. doi: 10.1055/s-0030-1255115. Epub 2010 Jul 19. PMID 20645233
- [Background] Silva AM, Fields DA, Heymsfield SB, Sardinha LB. Relationship between changes in total-body water and fluid distribution with maximal forearm strength in elite judo athletes. J Strength Cond Res. 2011 Sep;25(9):2488-95. doi: 10.1519/JSC.0b013e3181fb3dfb. PMID 21869630
- [Background] Silva AM, Matias CN, Santos DA, Rocha PM, Minderico CS, Sardinha LB. Increases in intracellular water explain strength and power improvements over a season. Int J Sports Med. 2014 Dec;35(13):1101-5. doi: 10.1055/s-0034-1371839. Epub 2014 Jul 10. PMID 25009970
- [Background] Armstrong LE. Assessing hydration status: the elusive gold standard. J Am Coll Nutr. 2007 Oct;26(5 Suppl):575S-584S. doi: 10.1080/07315724.2007.10719661. PMID 17921468
- [Background] Armstrong LE, Maughan RJ, Senay LC, Shirreffs SM. Limitations to the use of plasma osmolality as a hydration biomarker. Am J Clin Nutr. 2013 Aug;98(2):503-4. doi: 10.3945/ajcn.113.065466. No abstract available. PMID 23873679
- [Background] Barley OR, Chapman DW, Abbiss CR. Reviewing the current methods of assessing hydration in athletes. J Int Soc Sports Nutr. 2020 Oct 30;17(1):52. doi: 10.1186/s12970-020-00381-6. PMID 33126891
- [Background] Kyle UG, Bosaeus I, De Lorenzo AD, Deurenberg P, Elia M, Gomez JM, Heitmann BL, Kent-Smith L, Melchior JC, Pirlich M, Scharfetter H, Schols AM, Pichard C; Composition of the ESPEN Working Group. Bioelectrical impedance analysis--part I: review of principles and methods. Clin Nutr. 2004 Oct;23(5):1226-43. doi: 10.1016/j.clnu.2004.06.004. PMID 15380917
- [Background] Hetherington-Rauth M, Leu CG, Judice PB, Correia IR, Magalhaes JP, Sardinha LB. Whole body and regional phase angle as indicators of muscular performance in athletes. Eur J Sport Sci. 2021 Dec;21(12):1684-1692. doi: 10.1080/17461391.2020.1858971. Epub 2021 Jan 18. PMID 33280537
- [Background] Raman A, Schoeller DA, Subar AF, Troiano RP, Schatzkin A, Harris T, Bauer D, Bingham SA, Everhart JE, Newman AB, Tylavsky FA. Water turnover in 458 American adults 40-79 yr of age. Am J Physiol Renal Physiol. 2004 Feb;286(2):F394-401. doi: 10.1152/ajprenal.00295.2003. Epub 2003 Nov 4. PMID 14600032
- [Background] Stegeman D, Hermens H. Standards for surface electromyography: The European project Surface EMG for non-invasive assessment of muscles (SENIAM). Enschede: Roessingh Research and Development. 2007:108-12.
- [Background] Puga AM, Lopez-Oliva S, Trives C, Partearroyo T, Varela-Moreiras G. Effects of Drugs and Excipients on Hydration Status. Nutrients. 2019 Mar 20;11(3):669. doi: 10.3390/nu11030669. PMID 30897748
- [Derived] Francisco R, Jesus F, Nunes CL, Santos P, Alvim M, Campa F, Schoeller DA, Lukaski H, Mendonca GV, Sardinha LFCB, Silva AMLA. H2OAthletes study protocol: effects of hydration changes on neuromuscular function in athletes. Br J Nutr. 2024 May 14;131(9):1579-1590. doi: 10.1017/S0007114524000308. Epub 2024 Feb 1. PMID 38299306